CLINICAL TRIAL: NCT00788294
Title: Pharmacokinetics And Safety Of A Single Dose Subcutaneous Or Intravenous Administration Of Tanezumab In Healthy Volunteers: An Open-Label, Non-Randomized Phase 1 Study
Brief Title: Measure Exposure Of Tanezumab In Healthy Volunteers When Administering The Drug Subcutaneously
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4091013
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2009-07

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics tanezumab subcutaneous bioavailability intravenous Japanese subjects
MeSH Terms: interventions — tanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- 10 mg IV (Active Comparator)
  Interventions: Biological: tanezumab
- 5 mg SC (Active Comparator)
  Interventions: Biological: tanezumab
- 10 mg SC (Active Comparator)
  Interventions: Biological: tanezumab
- 19 mg SC (Active Comparator)
  Interventions: Biological: tanezumab

INTERVENTIONS:
Biological: tanezumab — Drug solution given intravenously only once at dose of 10 mg
  Arms: 10 mg IV
Biological: tanezumab — Drug solution given subcutaneously only once at dose of 5 mg.
  Arms: 5 mg SC
Biological: tanezumab — Drug solution given subcutaneously only once at dose of 10 mg.
  Arms: 10 mg SC
Biological: tanezumab — Drug solution given subcutaneously only once at dose of 19 mg.
  Arms: 19 mg SC

SUMMARY:
The hypothesis of this study is that subcutaneous administration of tanezumab results in lower drug exposure compared to intravenous administration of tanezumab.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* BMI of 18-30 kg/m2
* more than 50 kg bodyweight.

Exclusion Criteria:

* Pregnant
* exposure to biologic type drugs within the last 3 months
* history of allergic or anaphylactic reaction to a biologic drug
* use of tobacco- or nicotine containing products that is more than what is in 5 cigarettes per day
* excessive alcohol use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Subcutaneous bioavailability | 16 weeks
Injection site reactions | 16 weeks
Immunogenicity | 16 weeks

SECONDARY OUTCOMES:
Nerve growth factor levels | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Cypress, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091013&StudyName=Measure%20Exposure%20Of%20Tanezumab%20In%20Healthy%20Volunteers%20When%20Administering%20The%20Drug%20Subcutaneously